CLINICAL TRIAL: NCT05583071
Title: Pilot-trial of Methotrexate, Tafasitamab (Minjuvi®), Lenalidomide (Revlimid®) and Rituximab in Patients Ineligible for HCT-ASCT With Primary Central Nervous System Lymphoma (PCNSL)
Brief Title: Methotrexate, Tafasitamab, Lenalidomide and Rituximab in Patients With PCNSL
Acronym: MTR²
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Cologne (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Peter Borchmann, Trial Chairman, University of Cologne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uni-Köln-4968
Record Dates: First submitted 2022-08-02; First posted 2022-10-17 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-04

CONDITIONS: Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — tafasitamab; Lenalidomide; Rituximab; Methotrexate

STUDY DESIGN:
Intervention Model Description: single-arm, prospective, multicenter, single-stage phase-II trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- combination of Tafasitamab (Minjuvi®), Lenalidomide, Rituximab and Methotrexate (Experimental): All patients will receive tafasitamab (Minjuvi®) 12 mg/KG body weight and rituximab 375 mg/m² on days 0 and 5, followed by methotrexate 3,5 g/m² on day 1 as an intravenous infusion. Lenalidomide will be administered orally at 20 mg/day during the first cycle and at 25 mg/day during subsequent cycles on days 4-17 of each 21-day cycle for a total number of 4 cycles. The treatment duration per patient will be 84 days.
  Interventions: Drug: Tafasitamab; Drug: Lenalidomide; Drug: Rituximab; Drug: Methotrexate

INTERVENTIONS:
Drug: Tafasitamab — IV
Drug: Lenalidomide — Oral
Drug: Rituximab — IV
Drug: Methotrexate — IV

SUMMARY:
Pilot-trial of Methotrexate, Tafasitamab (Minjuvi®), Lenalidomide (Revlimid®) and Rituximab in patients ineligible for HCT-ASCT with Primary Central Nervous System Lymphoma (PCNSL)

DETAILED DESCRIPTION:
This is a single-arm, prospective, multicenter, single-stage phase-II trial for patients aged 18-69 years with ECOG PS ≥2 or ≥70 years with previously untreated PCNSL, who are not eligible for HCT-ASCT at investigators decision. This trial evaluates the CRR rate after at least 2 cycles of MTR2, the incidence and severity of adverse events, progression-free survival, and overall survival after one year.

It is planned to enroll eligible patients with PCNSL, i.e. who receive at least 2 cycles of the combination of rituximab, MTX and the IMPs tafasitamab and lenalidomide, over a one-year period. Follow-up will be conducted for 1 year within the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-69 years with ECOG PS ≥2 or age ≥70 years, and ineligible for HCT-ASCT as per investigators discretion
2. Previously untreated, histologically (or cytologically) confirmed diagnosis of primary B-cell lymphoma of the central nervous system (PCNSL) by local pathologist. Diagnostic sample obtained by stereotactic or surgical biopsy, CSF cytology examination or vitrectomy
3. At least one measurable lesion
4. Adequate organ function:

   * Adequate kidney function, defined as:

     * Serum creatinine estimated glomerular filtration rate (MDRD) ≥ 50 ml/min
   * Adequate hepatic function, defined as:

     * ALAT and ASAT ≤ 3 ULN
     * Bilirubin ≤ 2.0 mg/dl (except for Meulengracht disease)
   * Adequate bone marrow function, defined as:

     * White blood cell (WBC) count ≥ 3000/µL or absolute neutrophil count (ANC) ≥ 1000/µL
     * Platelets ≥ 50.000/µL
     * Hemoglobin > 8.0 g/dl
   * Adequate cardiac function, defined as:

     * Cardiac ejection fraction ≥ 40%
   * Adequate pulmonary function as per investigators discretion
5. Written, signed, and dated informed consent for the trial provided by the participant
6. Female persons are eligible to participate if they are post-menopausal or females of no childbearing potential or if they agree to use a method of contraception considered safe described in Section 12.1.2.1.
7. Male persons with female partners of childbearing potential are eligible to participate if they agree to contraceptive methods as described in Section 12.1.2.2.

Exclusion Criteria:

1. Prior treatment for PCNSL with the exception of a pre-phase treatment comprising steroid treatment and / or single application of rituximab 375 mg/m² and methotrexate 3.5 g/m²
2. Systemic lymphoma manifestation outside the CNS
3. Diagnosis of previous Non-Hodgkin lymphoma at any time
4. Primary vitreoretinal or leptomeningeal lymphoma without manifestation in the brain parenchyma or spinal cord
5. HIV infection of any stage as determined by presence of anti-HIV antibodies (confirmatory test) and / or presence of RNA confirmed by PCR
6. Previous or concurrent malignancies with the following exceptions:

   * Surgically cured carcinoma in-situ
   * Other kinds of cancer without evidence of disease for at least 5 years
7. Hypersensitivity to study treatment or any component of the formulation
8. Stomatitis or gastrointestinal ulcerations preventing the use of methotrexate
9. Hepatitis B, hepatitis C or hepatitis E infection as determined by PCR
10. Severe active infection
11. Congenital or acquired immunodeficiency including previous organ transplantation
12. Pregnant or nursing (lactating) women.
13. Lack of accountability and inability to appreciate the nature, meaning and consequences of the trial and to formulate their own wishes correspondingly
14. Non-compliance, for reasons including, but not limited to the following:

    1. Increased alcohol consumption, drug dependency or substance abuse that would interfere with cooperation with requirements of the trial
    2. Refusal of blood products during treatment
    3. Any similar circumstances that appear to make protocol treatment or long-term follow-up impossible
15. Relationship of dependence or employer-employee relationship to the sponsor or the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
complete response rate (CRR) | At the end of cycle 2 (each cycle is 21 days)
  The CRR will be determined by IRC and according to IPCG criteria. This endpoint reflects the proportion of patients who can potentially proceed to different consolidation or maintenance strategies to achieve durable responses.

SECONDARY OUTCOMES:
Best overall response rate (BORR) | At the end of cycle 4 (each cycle is 21 days)
  is defined as the rate of patients having achieved a CR or PR according to at least one post-baseline tumor assessment
Progression-free survival (PFS) | After 1 year
  will be calculated for each patient as time between the start of treatment with MTR2 and the date of first progression, relapse or death or, in cases of continuing response, the date of the last documented follow-up (FU-CRF or written medical report).
Overall survival (OS) | After 1 year
  will be calculated for each patient as time between the start of treatment with MTR2 and the date of death or the date of the last documented follow-up (FU-CRF or written medical report).
Incidence and severity of adverse events | during induction therapy
  Incidence and severity of adverse events, including toxic deaths during induction therapy will be summarized based on CTCAE grades

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (6):
  - Klinikum Stuttgart - Katharienenhospital, Stuttgart, Baden-Wurttemberg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Würtemberg
  - University of Cologne, Cologne, Germany
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg, Hamurg
  - Universitätsklinikum Essen, Essen, Nordrhein Westphalen
  - Charité - Universitätsmedizin Berlin, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: No